CLINICAL TRIAL: NCT03896035
Title: Improving Outcomes for Older Veterans With Chronic Back Pain and Depression (CDA 14-425)
Brief Title: Improving Outcomes for Older Veterans With Chronic Back Pain and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CDX 19-001; K2HX001916 (Other: VA HSRD)
Record Dates: First submitted 2019-02-05; First posted 2019-03-29 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-08

CONDITIONS: Chronic Back Pain; Depression; Aging
Keywords: Chronic Back Pain; Depression; Veterans; Aging
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This pilot RCT will use a waitlist control
Who Masked: Outcomes Assessor
Masking Description: The research staff conducting outcomes assessments will be blinded to whether the subject is in active or waitlist group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Waitlist Control Group (No Intervention): The waitlist control group will continue with management of chronic back pain and depression per usual care. All participants, regardless of what group they have been assigned to will undergo several outcome assessments (pre-screening, baseline, mid-point, final assessments) conducted by a blinded research assistant. Subjects randomized to the waitlist control group will be offered the same intervention once the active intervention group has completed the active sessions and assessments.
- Behavioral Intervention Group (Experimental): For participants assigned to the intervention arm, trained health coaches will deliver the intervention via telephone. All participants, regardless of what group they have been assigned to will undergo several outcome assessments (pre-screening, baseline, mid-point, final assessments) conducted by a blinded research assistant.
  Interventions: Behavioral: Behavioral Intervention Group

INTERVENTIONS:
Behavioral: Behavioral Intervention Group — The behavioral intervention is designed for older Veterans with cLBP and depression and will include 8 individual telephone sessions delivered by health coaches over a period of 10-20 weeks (up to 5 months total, accounting for additional time between sessions if needed).
  Arms: Behavioral Intervention Group

SUMMARY:
The overarching goal of this study is to develop and evaluate a telephone delivered behavioral change intervention for older Veterans with chronic low back pain (cLBP) and comorbid depression, and to ultimately assess its effect on cLBP-related pain, depressive symptoms, and disability.

Investigators will conduct a pilot randomized controlled trial to assess feasibility for older Veterans with cLBP and depression assigned to receive the behavioral interventions (n=25) versus waitlist control (n=25). For participants assigned to the intervention arm, trained health coaches will deliver the intervention via telephone. All participants, regardless of what group they have been assigned to will undergo several outcome assessments (pre-screening, baseline, mid-point, final assessments) conducted by a blinded research assistant. Subjects randomized to the waitlist control group will be offered the same intervention once the active intervention group has completed the active sessions and assessments.

DETAILED DESCRIPTION:
In this pilot RCT, investigators will assess the feasibility for older Veterans with cLBP and depression assigned to receive the behavioral intervention (n=25) versus the waitlist control (n=25). Follow-up will also include assessments at 6 months and 12 months post-intervention.

Overview of Proposed intervention: The behavioral intervention is designed for older Veterans with cLBP and depression and will include 8 individual telephone sessions delivered by health coaches over a period of 10-20 weeks (up to 5 months total, accounting for additional time between sessions if needed). Exceptions may be made for highly motivated subjects who had unfortunate life circumstances arise.

For the physical activity component of the intervention, investigators will provide an Omron pedometer to subjects, as previously used in VA research studies. The Omron pedometer will be set up by the research team (stride length, setting date/time) and will be mailed to the subject's home in between session 1 and 2. The health coach will remind the subject that this pedometer will arrive via United States Postal Service mail to their home and to call the research coordinator when it arrives. The research team will provide technical assistance and instructions to the subject regarding use of the Omron pedometer (to be worn on the waist band, daily, all day aside from showers/baths). The research team will also verbally show the subject how to press the mode and memory buttons to obtain weekly step counts for documentation/tracking physical activity. The subjects will be prompted by the health coach or research staff to report out weekly step counts during subsequent coaching sessions.

In addition to the assessments outlined later in this protocol, specifically at 12 months, investigators will conduct in-depth semi-structured interviews with ~10-15 participants (8 from both arms of the pilot trial, the health coaches, 2 primary care providers, and 1 mental health provider) using purposive sampling. The health coach/research coordinator will identify Veterans who are at higher risk for drop-out, were less engaged, or were particularly successful at achieving behavioral change. The purpose of this final interview is to learn about the barriers and facilitators to successful intervention delivery and participant retention from the Veteran, health coach, and provider perspective.

ELIGIBILITY:
Inclusion Criteria:

* Men and women Veterans aged 65+
* English-speaking
* Self-reported low back pain (+/-radiation) on most days for the past 3 months, that interferes with daily activities. Low back pain interferes with daily activities, assessed with the question "does your back pain limit your ability to do activities around the home or activities that you enjoy?"
* Chronic low back pain with intensity of 4 or higher on 10 point scale
* Depression, PHQ-9>10 stable (per chart review, no psychotic or suicidal ideation; confirmed over telephone)
* Capable of participating in home-based activity

Exclusion Criteria:

* No telephone
* Not English speaking
* Unwilling to be randomized to either study arm
* Self-reported uncorrected hearing or visual disturbance precluding ability to participate in telephone sessions or read pedometer screen
* Cognitive impairment, assessed by Memory Impairment Screen
* Lumbar surgery within the last year
* Self-reported dependence on wheelchair, bed-bound, or severe balance impairment (unable to participate in physical activity intervention)
* Illness requiring hospitalization within the last 3 months. Specific question: Have you been hospitalized for an illness in the past 3 months that would make participating in a physical activity program challenging or unsafe? (Examples include: fall, gout attacks, stroke, heart attack, heart failure, or surgery for blocked arteries)
* Suicidal ideation, prior psychotic episodes requiring hospitalization within the last year

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Una E. Makris, MD MSc, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (1):
- VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
Started | 24 | 26
Completed | 22 | 15
Not Completed | 2 | 11
Not completed — Lost to Follow-up | 2 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Health/family health issues during COVID | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Waitlist Control Group | Behavioral Intervention Group | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.21 (3.11) | 70.96 (3.49) | 71.08 (3.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 19 | 21 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 11 | 14 | 25
  Black, non-Hispanic | 11 | 10 | 21
  Hispanic, any race | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 26 | 50
Pain Scale [Mean (Standard Deviation); unit: units on a scale] — PEG-3 measures pain interference. Pain intensity on 0-10 scale where higher values are worse pain.
  units on a scale | 6.81 (1.78) | 6.76 (1.70) | 6.78 (1.72)
Depression [Mean (Standard Deviation); unit: units on a scale] — PHQ-9 measures depressive symptom severity. Scored between 0-27 with higher numbers indicated worse depression.
  units on a scale | 12.75 (4.78) | 13.92 (4.89) | 13.36 (4.82)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Intervention Completion
Description: Feasibility Outcome includes percentage of participants completing each arm
Time Frame: Through intervention delivery of 8 sessions, up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
Number analyzed (Participants) | 24 | 26
Participants | 22 | 15

2. Secondary Outcome: Pain Scale- PEG-3
Description: Pain intensity on 0-10 scale where higher values are worse pain; PEG-3 assesses 3 aspects of pain interference and averages these values
Time Frame: Through study completion, up to 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
Number analyzed (Participants) | 21 | 15
units on a scale | 6.57 (1.89) | 5.13 (2.04)

3. Secondary Outcome: Roland Morris Disability Questionnaire (RMDQ)
Description: Disability related to back pain. Scale ranges from 0-24 with larger numbers indicating worse disability related to chronic back pain
Time Frame: Through study completion, up to 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
Number analyzed (Participants) | 21 | 15
score on a scale | 17.10 (4.05) | 13.07 (4.22)

4. Secondary Outcome: Depression
Description: Depression: Patient Health Questionnaire (PHQ-9) scored between 0-27 with higher numbers indicated worse depression
Time Frame: Through study completion, up to 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
Number analyzed (Participants) | 21 | 15
score on a scale | 10 (4.35) | 7.4 (4.90)

ADVERSE EVENTS:
Time Frame: Adverse event data reported over 1 year period
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

LIMITATIONS AND CAVEATS:
This pilot trial was designed to assess feasibility: ability to recruit, refine protocols and procedures and retain participants. The pilot trial was active during 2019-2020 when COVID restrictions were severe, locally, and several participants in the active arm were lost to follow-up for health related reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT03896035/Prot_SAP_000.pdf